CLINICAL TRIAL: NCT03196648
Title: A Randomized Trial Evaluating the Efficacy of a Gum Health Formulation on Gingival Inflammation, Oral Malodor and Tooth Whitening
Brief Title: Randomized Trial of a Gum Health Formulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glo Science, Inc. (Industry)
Collaborators: The Forsyth Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLO-002
Record Dates: First submitted 2017-06-19; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Periodontal Diseases; Gingivitis; Periodontitis; Halitosis
Keywords: Gingivitis; Periodontal disease; Inflammation; Teeth whitening; Breath freshening; Periodontal pathogens; Bleeding on probing
MeSH Terms: conditions — Periodontal Diseases; Gingivitis; Periodontitis; Halitosis; Inflammation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gingival health formulation in accelerating device (Experimental): The interventional gingival health formulation is applied to the participant's mouth by means of an intra-oral accelerating device for a single eight-minute application, daily. Participants were instructed to brush their teeth with an OTC toothpaste twice daily, morning and night.
  Interventions: Other: Gingival health formulation in an accelerating device; Other: OTC fluoride toothpaste
- Gingival health formulation on a toothbrush (Experimental): The interventional gingival health formulation is applied to the participant's mouth by means of a toothbrush and OTC toothpaste, together with the formulation in equal amounts, for two-minute applications twice daily, morning and night.
  Interventions: Other: Gingival health formulation on a toothbrush; Other: OTC fluoride toothpaste
- Control group (Split mouth design) (Active Comparator): The control group did not receive the interventional gingival health formulation. Participants were instructed to brush their teeth with a toothbrush and OTC toothpaste twice daily, morning and night. In addition, participants were instructed to floss only half of their mouth daily, having the non-flossed half serve as an untreated comparative control of toothbrushing alone.
  Interventions: Other: OTC fluoride toothpaste

INTERVENTIONS:
Other: Gingival health formulation in an accelerating device — The intervention is a gingival health formulation for soft tissue maintenance, oral malodor and gentle teeth whitening to be used with the GLO Science Device
  Other Names: ECO Balance; GLO Science accelerating device
  Arms: Gingival health formulation in accelerating device
Other: Gingival health formulation on a toothbrush — The intervention is a gingival health formulation for soft tissue maintenance, oral malodor and gentle teeth whitening to be used on a toothbrush together with toothpaste.
  Other Names: ECO Balance
  Arms: Gingival health formulation on a toothbrush
Other: OTC fluoride toothpaste — OTC anti-cavity toothpaste containing fluoride and sodium monofluorophosphate.
  Other Names: GLO Science Antioxidant Toothpaste

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a newly formulated foaming gel product on gingivitis and/or moderate periodontitis when used with or without the GLO Science accelerating device (GLO Device), compared to standard tooth brushing with antioxidant whitening toothpaste with or without flossing (split mouth design for control group).

This is a 60-day randomized single blinded parallel group study. After 42 days, all use of interventional products were discontinued, and the participants returned to the clinical center at day 60 for final measurements. The primary outcomes assessed in this study were the differences in gingival index (GI) and bleeding on probing (BOP) from baseline to 42 & 60 days. The secondary outcomes are tooth whitening, oral malodor, pocket depth and plaque amount.

It is hypothesized that participants using the gingival health product with the GLO Device will experience greater reductions in GI & BOP measurements than the control group, as well as participants using the gingival health product on a toothbrush alone.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to read, understand and sign an Informed Consent Form
* Good general health as evidenced by the medical history
* Between 18 and 55 years of age
* Male or female
* Minimum of 20 teeth, excluding crowns and third molar teeth
* Mean whole mouth Gingival Index >/=2.0 at baseline; sites with </=7mm pocket depth
* Willing to abstain from all oral hygiene procedures 12-18 hours prior to clinical visits
* Willing to abstain from eating and drinking for 2 hours prior to clinical visits, only drinking water is allowed
* Willing to abstain from chewing gums, oral whitening products, mouthwashes and tobacco products for the study duration
* Able to understand and follow study directions

Exclusion Criteria:

* Chronic use of photosensitizing medications including NSAIDs, antidepressants, antibiotics and beta-blockers
* Diagnosed with diabetes
* Presence of orthodontic appliances
* Presence of large restorations, crown or veneer at the anterior of both upper and lower teeth (including premolar teeth)
* A soft or hard tissue tumor of the oral cavity
* Carious lesions requiring immediate treatment
* Patients with severe internal (tetracycline stains) and external discoloration (fluorosis)
* Patients with severe chronic periodontitis, aggressive periodontitis, acute necrotizing ulcerative gingivitis, or generalized gingival recession >2mm as evidenced by clinical oral exam
* Pregnant or breast-feeding women
* Allergy to home bleaching products such as hydrogen peroxide and carbide peroxide
* Use of antibiotics within 3 months of enrollment
* History of drug use that is associated with gum overgrowth (i.e., Dilantin, nifedipine, etc.)
* Chronic use of medication such as steroids, anti-coagulant medications, immunosuppressant medication or any other medications or medical conditions that in the opinion of the Investigator would interfere with the evaluation or confound interpretation of the study results. Use of low dose of ASA (<325mg) is permitted.
* Medical condition which requires pre-medication prior to dental visits/procedures
* Current smoking and former smoking within one year of enrollment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Differences in bleeding on probing | Baseline to 42 days
Differences in Gingival Index | Baseline to 42 days

SECONDARY OUTCOMES:
Difference in Plaque Index | Baseline to 42 days
Difference in mean probing depth | Baseline to 42 days
Change in oral malodor | Baseline to 42 days
  Chromatographic measure of volatile sulfur compounds (hydrogen sulfide, dimethyl sulfide, methyl mercaptan)
Change in tooth whitening | Baseline to 42 days
Change in sub-gingival bacterial profile | Baseline to 28 days
  DNA-DNA Hybridization Checkerboard; Measurement of bacterial load
Change in inflammatory cytokines | Baseline to 28 days
  Measurement of IL-1B, TNF-a, IL-6, IL-8 & MCP-1 volume from gingival crevicular fluid samples

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Hasturk, DDS, PhD, Principal Investigator — The Forsyth Institute
Locations (1):
- The Forsyth Institute, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No